CLINICAL TRIAL: NCT03489772
Title: A Randomized, Placebo-Controlled, Double-Blind Study of Escalating Single Doses of ITI-214 in Healthy Volunteers to Determine Central Nervous System Engagement, Safety and Tolerability
Brief Title: Study of ITI-214 in Healthy Volunteers to Determine CNS Engagement
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Collaborators: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: ITI-214-106
Record Dates: First submitted 2018-03-09; First posted 2018-04-05 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — ITI-214

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 1 mg ITI-214 (Experimental): Single dose
  Interventions: Drug: ITI-214
- 10 mg ITI-214 (Experimental): Single dose
  Interventions: Drug: ITI-214
- Placebo (Placebo Comparator): Single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ITI-214 — Oral
  Arms: 1 mg ITI-214; 10 mg ITI-214
Drug: Placebo — Oral
  Arms: Placebo

SUMMARY:
This is a single site, randomized, double-blind, placebo-controlled, within-subjects study design in healthy volunteers. Escalating single doses of ITI-214 will be evaluated using functional magnetic resonance imaging (fMRI) to determine central nervous system engagement. Safety and tolerability also will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female, 18 - 45 years
* Fluent and literate in English and able to provide written informed consent
* BMI between 18.5 and 38.0 kg/m2 and minimum body weight of 50 kg

Exclusion Criteria:

* Recent exposure to any investigational product
* Previous exposure to relevant fMRI task(s)
* Considered medically unsuitable for participation
* Has any contraindication for BOLD fMRI

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-08-05 (Actual)

PRIMARY OUTCOMES:
BOLD MRI signals in the anterior insula during the extinction phase of a Fear Conditioning task | 1-3 hours post-dose
  Changes in brain activation
BOLD MRI signals in the inferior frontal gyrus during the Stop Signal Task | 1-3 hours post-dose
  Changes in brain activation

SECONDARY OUTCOMES:
BOLD fMRI signals elicited by fear conditioning stimulus | 1-3 hours post-dose
  Changes in brain activation in amygdala, prefrontal cortex, and/or insula cortex
BOLD fMRI signals elicited by the Stop versus Go signal | 1-3 hours post-dose
  Changes in brain activation in dorsolateral prefrontal cortex and/or anterior cingulate cortex
Number of subjects with reported or observed treatment-related adverse events | 0-5 hours post-dose
  Safety and tolerability

OTHER OUTCOMES:
BOLD fMRI signals elicited in the amygdala, insula and medial prefrontal cortex | 1-3 hours post-dose
  Pharmacodynamics

CONTACTS AND LOCATIONS:
Overall Officials: Robert Davis, PhD, Study Director — Intra-Cellular Therapies, Inc.
Locations (1):
- Laureate Institute for Brain Research, Inc., Tulsa, Oklahoma, United States

REFERENCES:
- [Derived] Khalsa SS, Victor TA, Kuplicki R, Yeh HW, Vanover KE, Paulus MP, Davis RE. Single doses of a highly selective inhibitor of phosphodiesterase 1 (lenrispodun) in healthy volunteers: a randomized pharmaco-fMRI clinical trial. Neuropsychopharmacology. 2022 Sep;47(10):1844-1853. doi: 10.1038/s41386-022-01331-3. Epub 2022 Apr 29. PMID 35488084